CLINICAL TRIAL: NCT06327126
Title: Efficacy and Safety of Single-session Endoscopic Stone Extraction for Treating Acute Cholangitis Accompanied With Choledocholithiasis
Brief Title: Efficacy and Safety of Single-session Endoscopic Stone Extraction
Status: Completed | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BFHHZS20240001
Record Dates: First submitted 2024-03-11; First posted 2024-03-25 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-03

CONDITIONS: Choledocholithiasis With Acute Cholangitis
Keywords: Choledocholithiasis; Acute Cholangitis; Endoscopic Retrograde Cholangiopancreatography
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- two-session treatment group: two-session ERCP
  Interventions: Procedure: two-session ERCP
- single-session treatment group: single-session ERCP
  Interventions: Procedure: single-session ERCP

INTERVENTIONS:
Procedure: two-session ERCP — early endoscopic drainage followed by endoscopic stone extraction
  Groups: two-session treatment group
Procedure: single-session ERCP — directly endoscopic stone extraction
  Groups: single-session treatment group

SUMMARY:
This is a retrospective study, including approximately 600 patients with acute cholangitis accompanied with choledocholithiasis, who treated with single-session or two-session endoscopic stone extraction at Beijing friendship hospital. The investigators assessed the outcomes of single-stage and two-stage endoscopic stone extraction.

DETAILED DESCRIPTION:
Acute cholangitis is an acute inflammation caused by obstruction of the bile duct, of which choledocholithiasis is the most common cause. Without timely removal of the obstruction or control of the infection, cholangitis can get worse and even become life-threatening. Therefore, timely and effective treatment is essential for patients with acute cholangitis combined with choledocholithiasis. Endoscopic retrograde cholangiography (ERCP) is used as the first-line treatment for choledocholithiasis-associated acute cholangitis. Previous guidelines recommended two-session endoscopic therapy. Endoscopic biliary drainage as the initial treatment, followed by endoscopic stone extraction after cholangitis improved. In recent years, studies have found that single-session endoscopic stone extraction is safe and effective for patients without serious organ function impairment. Meanwhile, single-session endoscopic lithotomy can avoid the second ERCP intervention, which can relieve the pain of patients, reduce medical costs and shorten the length of hospital stay. However, there is still insufficient evidence on the effectiveness and safety of early single-session ERCP lithotomy. The aim of this study is to evaluate the efficacy and safety of single-session endoscopic stone extraction for acute cholangitis associated with choledocholithiasis, so as to provide reference of clinical treatment.

In a retrospective analysis, approximately 600 patients with acute cholangitis accompanied with choledocholithiasis, who treated with single-session or two-session endoscopic stone extraction at Beijing friendship hospital were studied. The investigators assessed the outcomes of single-stage and two-stage endoscopic stone extraction.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Patients met the Tokyo Guidelines 2018 (TG18) diagnosis of acute cholangitis
3. Imaging examination confirmed the presence of choledocholithiasis
4. Patients received endoscopic single-session stone extraction or two-session treatment involving stone removal after drainage

Exclusion Criteria:

1. Common bile duct with benign or malignant stenosis
2. Changes in the anatomical structure of the stomach or duodenum
3. Patients complicated with severe acute pancreatitis
4. Patients who underwent endoscopic intervention before admission
5. Patients received percutaneous transhepatic cholangio drainage (PTCD) or other invasive interventions besides endoscopic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed with acute cholangitis associated with choledocholithiasis underwent single-session stone extraction or two-session treatment involving stone removal after drainage at Beijing Friendship Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Success rate of complete stone removal | during the operation
  Segmental angiography was performed by balloon closure to determine the presence or absence of negative stone shadow
ERCP-related complication rate | from the operation to 1 month after the operation
  The complications include pancreatitis, hemorrhage, perforation, pneumonia, etc. The results of intraoperative endoscopic observation, postoperative symptoms and signs, blood routine examination, amylase, lipase, and imaging and endoscopic examination were measured.

SECONDARY OUTCOMES:
Length of stay | perioperatively
  Total time from admission to discharge.
Hospital expenses | perioperatively
  Total expenses from admission to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Fujing Lv, M.D., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No